CLINICAL TRIAL: NCT06588959
Title: "Validity and Reliability of the 6-minute Pegboard Ring Test in Patients with Scleroderma
Brief Title: 6-minute Pegboard Ring Test in Patients with Scleroderma
Status: Not yet recruiting | Type: Observational
Sponsor: Yasemin GEDIKLI (Other)
Collaborators: Scientific Research Projects (Unknown)
Responsible Party: Sponsor-Investigator, Yasemin GEDIKLI, Faculty of Health Sciences Physiotherapy and Rehabilitation- Research assistant, Selcuk University
Organization: Selcuk University (Other)
Other Study IDs: SelcukU-FTR-YG-01
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Systemic Sclerosis (SSc); Scleroderma
Keywords: Exercise Test, Upper Extremity, arm exercise endurance
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with systemic sclerosis
  Interventions: Other: validity and reliability study

INTERVENTIONS:
Other: validity and reliability study — Determination of strength, endurance and exercise capacity of the upper extremities is an important issue in scleroderma management. 6PBRT, which is one of the tests serving this purpose, has been found to be valid and reliable in patients with chronic obstructive pulmonary disease and asthma, but when the literature is reviewed, it is seen that 6PBRT has not been studied in patients with scleroderma. This study was planned as a non-interventional safety study. The study will investigate the validity and reliability of 6PBRT in patients with scleroderma. In this context, the test will be performed 2 times with a 1-hour rest break. Dyspnea and fatigue will be assessed using the Borg scale and muscle oxygenation, heart rate and blood pressure will be recorded before and after 6PBRT. The level of dyspnea and fatigue and baseline values of heart rate will be checked before the second trial to ensure patients are stable. All assessments will be performed by the same physiotherapist.

SUMMARY:
The aim of this observational study was to evaluate the reliability and validity of the 6-minute pegboard and ring test (6PBRT) in patients with systemic sclerosis. The main question it aims to answer is:

- Is 6PBRT a valid and reliable method to assess upper extremity functional capacity in patients with systemic sclerosis? Participants will repeat the 6PBRT 2 times 1 hour apart. In addition, respiratory muscle strength (MIP-MEP), upper extremity muscle strength (hand dynanometer and hand-held dynanometer), muscle oxygen saturation (Moxy Monitor Device) will be evaluated.

DETAILED DESCRIPTION:
Upper extremity functions are of great importance, especially activities of daily living. There are opinions that the impairment of the upper extremity in scleroderma is greater than that of the lower extremity and affects the functional status of individuals more. This activity limitation is related to many activities of daily living, including unsupported upper limb movements that lead to dyspnea and fatigue in patients with cardiopulmonary disease. Therefore, determining the strength, endurance and exercise capacity of the upper extremities is an important issue in scleroderma management. One of the tests that serves this purpose is the 6PBRT, which has been found to be valid and reliable in patients with chronic obstructive pulmonary disease and asthma.

It was planned as a non-interventional reliability study. The study will investigate the validity and reliability of 6PBRT in patients with scleroderma. In this context, a 1-hour rest break will be given after the first test. Dyspnea and fatigue will be assessed using the Borg scale and muscle oxygenation, heart rate and blood pressure will be recorded before and after 6PBRT. After the 1-hour rest period, the second trial of 6PBRT will be performed. The level of dyspnea and fatigue and initial values of heart rate will be checked before the second trial to ensure that patients are stable. All assessments will be performed by the same physiotherapist. In addition, participants will be assessed for respiratory muscle strength, upper limb muscle strength and muscle oxidation during the performance test.

The smallest sample size of the study was 40 subjects with a correlation coefficient of 0.95 between the two tests and 90% power at 95% confidence interval. 50 subjects are aimed to be recruited against a 20% drop-out risk. Shapiro-Wilk test and histogram plots will be used to check the normality of the data. Demographic and clinical characteristics of the participants will be reported using descriptive statistics. Two-way random effects and absolute agreement methods and intraclass correlation coefficient (ICC) will be used to assess test-retest reliability. Reliability strength will be interpreted as excellent for an ICC value >0.90. The 95% Confidence Interval (95% CI) will be calculated to investigate measurement variability.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-75
* 2013 To be diagnosed with systemic sclerosis according to ACR/EULAR classification criteria
* Being clinically stable
* Ability to adapt to tests (visual, cognitive, cooperative)

Exclusion Criteria:

* Those with neurological and/or musculoskeletal problems that may affect the work
* Presence of severe joint contracture or painful ulcers that may affect muscle strength measurement and walking
* Presence of severe infection or sepsis
* Being diagnosed with a known additional rheumatologic disease
* Any stage of cancer
* Pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at Selçuk University, Faculty of Health Sciences. The study will include volunteer individuals with systemic sclerosis who are eligible to participate in the study and who are being followed up and treated with a diagnosis of scleroderma in the Department of Rheumatology.
  -- Purposive sampling
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
6-Minute Pegboard and Ring Test | baseline
  It is used to assess upper extremity exercise capacity.The 6PBRT will be performed using a pegboard with two upper and lower pegs placed at and above the participants' shoulder level (20 cm). During the test, participants will use both hands simultaneously to move 10 lightweight wooden rings from the lower pegs to the upper pegs. Then, they will move the rings from the top pegs back to the bottom pegs. This activity will continue for six minutes. The aim is to move as many rings as possible during the six minutes. The score will be reported as the number of rings moved simultaneously. Every minute participants will be given standardized verbal encouragement. Heart rate, blood pressure, respiratory frequency, dyspnea and fatigue will be evaluated according to the Modified Borg Scale before and after the test.

SECONDARY OUTCOMES:
Demographic and Clinical Data | baseline
  Information on age, height, body weight, body mass index, gender, educational status, occupation, medication use, exercise habits and disease will be evaluated.
Extremity Muscle Strength Measurement | baseline
  Hand grip, elbow flexion, shoulder flexion and abduction muscle forces will be measured with a dynamometer.
Respiratory muscle strength measurement | baseline
  Intraoral pressure will be measured with a measuring instrument. They are easily applicable and simple measurements. Maximal voluntary inspiratory and expiratory pressures (MIP and MEP) are the most commonly used noninvasive method to measure respiratory muscle strength. It is based on Müller (maximal inspiration) and Valsalva (maximal expiration).
Muscle Oxygen Saturation | baseline
  Participants upper extremity muscle oxygen saturation will be assessed during 6PBRT.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhan S, Cerny FJ, Gibbons WJ, Mador MJ, Wu YW. Development of an unsupported arm exercise test in patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2006 May-Jun;26(3):180-7; discussion 188-90. doi: 10.1097/00008483-200605000-00013. PMID 16738459
- [Background] de Oliveira NC, Portes LA, Pettersson H, Alexanderson H, Bostrom C. Aerobic and resistance exercise in systemic sclerosis: State of the art. Musculoskeletal Care. 2017 Dec;15(4):316-323. doi: 10.1002/msc.1185. Epub 2017 Apr 5. PMID 28378937
- [Background] Calik-Kutukcu E, Tekerlek H, Bozdemir-Ozel C, Karaduz BN, Cakmak A, Inal-Ince D, Saglam M, Vardar-Yagli N, Sonbahar-Ulu H, Firat M, Arikan H, Kaya SB, Karakaya G. Validity and reliability of 6-minute pegboard and ring test in patients with asthma. J Asthma. 2022 Jul;59(7):1387-1395. doi: 10.1080/02770903.2021.1930040. Epub 2021 May 31. PMID 33985406
- [Background] Calderon LM, Pope JE. Scleroderma epidemiology update. Curr Opin Rheumatol. 2021 Mar 1;33(2):122-127. doi: 10.1097/BOR.0000000000000785. PMID 33481429
- [Background] Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996 Mar;76(3):248-59. doi: 10.1093/ptj/76.3.248. PMID 8602410
- [Background] Alkotob ML, Soltani P, Sheatt MA, Katsetos MC, Rothfield N, Hager WD, Foley RJ, Silverman DI. Reduced exercise capacity and stress-induced pulmonary hypertension in patients with scleroderma. Chest. 2006 Jul;130(1):176-81. doi: 10.1378/chest.130.1.176. PMID 16840399
- [Background] Ozsoy I, Ozcan Kahraman B, Ozsoy G, Ilcin N, Kahraman T, Acar S, Tekin N, Savci S. Determinants of the 6-minute pegboard and ring test as an unsupported upper-extremity exercise capacity measure in older adults with chronic obstructive pulmonary disease. Eur Geriatr Med. 2018 Dec;9(6):863-870. doi: 10.1007/s41999-018-0111-x. Epub 2018 Sep 25. PMID 34674474
- [Background] Chen YT, Kruger G, Devine A, Khanna D, Murphy SL. Experiences of Exergaming for Upper Extremity Exercises in People With Systemic Sclerosis. OTJR (Thorofare N J). 2023 Oct;43(4):665-675. doi: 10.1177/15394492231172934. Epub 2023 May 10. PMID 37162267
- [Background] Özcan Kahraman B, Özsoy İ, Tanrıverdi A, Akdeniz B, Özpelit E, Şentürk B, Acar S, Sevinç C, Savcı S. VALIDITY AND RELIABILITY OF THE 6-MINUTE PEGBOARD RING TEST IN PATIENTS WITH PULMONARY HYPERTENSION. Turk J Physiother Rehabil. 2020;31(2):210-7.